CLINICAL TRIAL: NCT02050282
Title: Prehospital Triage of Patients With Severe Dyspnea Using Point-of-Care N-terminal Pro-Brain Natriuretic Peptide. PreBNP Trial.
Brief Title: Prehospital Triage of Patients With Severe Shortness of Breath Using Biomarkers
Acronym: PreBNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Morten Thingemann Bøtker, MD, PhD student, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AU-PHAD01
Record Dates: First submitted 2014-01-23; First posted 2014-01-30 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Dyspnea
Keywords: Dyspnea; Prehospital; Biomarker; Heart failure; Triage; Randomized, controlled study
MeSH Terms: conditions — Dyspnea; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Business as usual (No Intervention): Triage and treatment based on routine clinical assessment as usual
- Supplementary NT-proBNP measurement (Experimental): Triage and treatment based on routine clinical assessment supplemented with measurement of NT-proBNP
  Interventions: Other: Supplementary NT-proBNP measurement

INTERVENTIONS:
Other: Supplementary NT-proBNP measurement — In patients randomized to the strategy with supplementary measurement of NT-proBNP, a blood sample will be drawn from the peripheral venous catheter that is routinely inserted and analyzed immediately using a COBAS H232 and Roche Diagnostics NT-proBNP assay.
  Arms: Supplementary NT-proBNP measurement

SUMMARY:
Breathlessness is a dangerous symptom. Preliminary data from national and regional Danish databases show, that patients with shortness of breath in the ambulance have a very high mortality. Breathlessness can be caused by many different conditions - but heart diseases and lung diseases are dominant. The mortality is especially high in patients with breathlessness caused by heart disease.

Distinguishing these different causes of breathlessness is a classical, often difficult, discipline in medicine. Visitation and guidance of treatment in patients with breathlessness in the prehospital setting relies on medical history and physical examination and as a consequence prehospital treatment for breathlessness is often non-specific. The use of heart-failure specific biomarkers may improve prehospital visitation and treatment of patients with breathlessness.

We hypothesize, that

1. Supplementing the routine examination by prehospital anesthesiologist with measurement of a biomarker for heart failure increases the proportion of patients with severe shortness of breath caused by heart disease triaged directly to department of cardiology
2. This strategy does not increase the proportion of patients with severe shortness of breath caused by non-heart disease triaged directly to department of cardiology

DETAILED DESCRIPTION:
Measurement of the biomarker for heart failure N-terminal pro-Brain Natriuretic Peptide (NT-proBNP):

In patients randomized to the strategy with supplementary measurement of NT-proBNP, a blood sample will be drawn from the peripheral venous catheter that is routinely inserted. This will be analyzed point-of-care in the ambulance.

Interpretation of NT-proBNP:

Cut-off values based on bootstrap-validated optimal cut-points for heart failure on will be used.

Confirmatory ('rule in') cut point

< 50 years: 450 pg/mL

50-75 years: 900 pg/mL

> 75 years: 1800 pg/mL

Exclusionary ('rule out') cut point

All patients: 300 pg/mL

The emergency physicians will be thoroughly informed about these cut-points, but told not to triage to department of cardiology or other department strictly according to NT-proBNP, but according to clinical assessment AND NT-proBNP.

ELIGIBILITY:
Inclusion Criteria:

All patients requiring dispatch of emergency physician because of severe dyspnea.

Severe dyspnea is defined by dyspnea plus at least ONE of the following

* Respiration frequency > 20 or < 8
* Saturation < 96 without supplementary oxygen
* Heart rate > 100 or < 50
* Systolic blood pressure < 100 or > 200
* Difficulty talking
* Central or peripheral cyanosis
* Use of accessory muscles of respiration
* Glasgow coma scale score < 15

AND because of the physical condition, the patient is not able to give informed consent

Exclusion Criteria Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with dyspnea caused by heart disease initially triaged to department of cardiology | Within 1 day from randomization
  An endpoint committee determines final diagnoses as "dyspnea caused by heart disease", "dyspnea caused by lung disease" and "dyspnea caused by other diseases" based on clinical and paraclinical data excluding prehospital NT-pro-BNP value

SECONDARY OUTCOMES:
Proportion of patients with dyspnea of other etiologies initially triaged to department of cardiology | Within 1 day from randomization
  An endpoint committee determines final diagnoses as "dyspnea of cardiac origin" and "dyspnea of non-cardiac origin" based on clinical and paraclinical data excluding prehospital NT-pro-BNP value
Proportion of patients with dyspnea caused by heart disease that receives pulmonary medication | Within 1 day
  beta2-agonist inhalations, combined ipratropium/b2-agonist inhalations, intravenous b2-agonists, intravenous corticosteroids
Length of hospital stay | Up to three months from randomization
  Time from hospital admission related to the inclusion event to discharge from hospital
Intensive care unit admission rate | Up to three months from randomization
  Within the time from hospital admission related to the inclusion event to discharge from hospital related to inclusion event
All-cause re-admission | Within 3 months of randomization
Proportion of patients not admitted to hospital | Within 24 hours
  Proportion of patients not admitted to hospital in relation to the inclusion event
All-cause mortality | Within 30 days of randomization
Proportion of patients with dyspnea caused by lung disease, that receives traditional heart failure medication | Within 1 day
  Loop diuretics, nitrates, opiates
Proportion of patients with correct diagnosis of congestive heart failure in the prehospital setting | Within 1 day of randomization
  An endpoint committee determines final diagnoses based on clinical and paraclinical data excluding prehospital NT-pro-BNP value
Proportion of patients where congestive heart failure is correctly disproved in the prehospital setting | Within 1 day of randomization
  An endpoint committee determines final diagnoses based on clinical and paraclinical data excluding prehospital NT-pro-BNP value

CONTACTS AND LOCATIONS:
Overall Officials: Morten Thingemann Bøtker, MD, Principal Investigator — Central Denmark Region; Christian Juhl Terkelsen, MD, DmSc, Study Director — Department of Cardiology B, Aarhus University Hospital, Skejby, Denmark; Hans Kirkegaard, Professor, Study Chair — Aarhus University Hospital; Erika Frischknecht Christensen, MD, Study Chair — Central Denmark Region; Thorbjørn Grøfte, MD, PhD, Study Chair — Central Denmark Region; Carsten Stengaard, MD, PhD, Study Chair — Department of Cardiology B, Aarhus University Hospital, Skejby, Denmark
Locations (9):
- Denmark (9):
  - Critical Care Team Aarhus, Prehospital Emergency Medical Services, Aarhus, Central Jutland
  - Critical Care Team Grenaa, Prehospital Emergency Medical Services, Grenå, Central Jutland
  - Critical Care Team Herning, Prehospital Emergency Medical Services, Herning, Central Jutland
  - Critical Care Team Holstebro, Holstebro, Central Jutland
  - Critical Care Team Horsens, Prehospital Emergency Medical Services, Horsens, Central Jutland
  - Critical Care Team, Lemvig, Prehospital Emergency Medical Services, Lemvig, Central Jutland
  - Critical Care Team Randers, Prehospital Emergency Medical Services, Randers, Central Jutland
  - Critical Care Team Silkeborg, Prehospital Emergency Medical Services, Silkeborg, Central Jutland
  - Critical Care Team, Viborg, Prehospital Emergency Medical Services, Viborg, Central Jutland

REFERENCES:
- [Derived] Botker MT, Jorgensen MT, Stengaard C, Seidenfaden SC, Tarpgaard M, Granfeldt A, Mortensen TO, Grofte T, Friesgaard KD, Maerkedahl R, Pedersen AB, Lundorff S, Hansen TM, Kirkegaard H, Christensen EF, Terkelsen CJ. Prehospital triage of patients suffering severe dyspnoea using N-terminal pro-brain natriuretic peptide, the PreBNP trial: a randomised controlled clinical trial. Eur Heart J Acute Cardiovasc Care. 2018 Jun;7(4):302-310. doi: 10.1177/2048872617709985. Epub 2017 May 11. PMID 28492084